CLINICAL TRIAL: NCT03065738
Title: Effect Of Reduction Osteotomy On Gap Balancing During Total Knee Replacement For Severe Varus Deformity
Brief Title: Effect of RO On GB During TKR Severe Varus Deformity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser E khalifa, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Alaa Safwat Taha
Record Dates: First submitted 2017-01-31; First posted 2017-02-28 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Genu Varum; Knee Osteoarthritis
Keywords: reduction osteotomy; knee arthroplasty
MeSH Terms: conditions — Genu Varum; Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osteoarthritis knee ,severe varus deformity (Experimental): reduction osteotomy in total knee replacement
  Interventions: Other: tibial reduction osteotomy in total knee replacement

INTERVENTIONS:
Other: tibial reduction osteotomy in total knee replacement — reduction osteotomy :downsizing of tibial tray with lateralization

SUMMARY:
Effect Of Reduction Osteotomy On Gap Balancing During Total Knee Replacement For Severe Varus Deformity

DETAILED DESCRIPTION:
Severe varus deformity with a tibio femoral angle of 15° or more as measured on full-length weight-bearing radiographs necessitates extensive release of the medial structures to gain neutral limb alignment during total knee arthroplasty (TKA). progressive releases of the medial structures are performed until medial and lateral envelopes are equally balanced. This technique, however, faces a risk of over-release and subsequent instability, ultimately resulting in the use of a thicker polyethylene insert or even a constrained-type prosthesis. Reduction osteotomy is known as a soft tissue-sparing technique for soft tissue balancing, and it is capable of reducing the amount of release required to balance the knee and of preventing over release of medial structures. Dixon et al . and Mullaji et al . proposed the effectiveness of down-sizing the tibial component in the case of knees with severe varus deformity Aim of the work: Assess the effect of reduction osteotomy on gab balancing during total knee arthroplasty for severe varus deformity -What is the amount of deformity correction achieved with reduction osteotomy during TKA in varus knees? - What is the correlation of amount of deformity correction achieved to the amount of bone osteotomized and the degree of varus deformity?

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe varus deformity more than 15 degrees (long film-mechanical axis)
* Patients with bone defect of medial tibial condyle

Exclusion Criteria:

* Patients with extra-articular deformity
* Patients with valgus deformity

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
HKA angle | immediate post operative
  standing A.P radiograph

SECONDARY OUTCOMES:
functional outcome by knee society score | one year follow up
  by knee society score

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Bakr, MD, Study Director — Assiut University
Locations (1):
- Assiut University School of medicine Vice Dean for Research and Post-Graduate Studies, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided